CLINICAL TRIAL: NCT02139891
Title: Randomized, Crossover Study of the Effects of MultiPoint Left Ventricular Pacing on Neurohormonal Activation.
Brief Title: Effects of Multipoint Pacing CRT-D on Neurohormonal Activation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Giovanni B Forleo, MD, PhD., University of Rome Tor Vergata
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PTVCARDIO022014
Record Dates: First submitted 2014-05-12; First posted 2014-05-15 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Heart Failure
Keywords: Cardiac Resynchronization Therapy; non responders; MultiPoint Pacing (MPP)
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MultiPoint Pacing "On" (Experimental): Patients will be randomized to the MPP-ON Arm vs MPP-OFF in in crossover fashion with 3 months in each period.
  Interventions: Device: Cardiac Resynchronization Therapy with MultiPoint Pacing
- MultiPoint Pacing "Off" (Active Comparator): Patients will be randomized to the MPP-OFF arm vs MPP-ON in crossover fashion with 3 months in each period.
  Interventions: Device: Cardiac Resynchronization Therapy with MultiPoint Pacing

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy with MultiPoint Pacing

SUMMARY:
This study will examine the additional clinical benefit conferred by multipoint pacing (MPP) compared to standard CRT over a period of 3 months. Patients will be randomized to MPP ON vs. OFF and followed for a total of 6 months. This includes two crossover periods for each pacing modality (MPP on vs. off).

DETAILED DESCRIPTION:
Cardiac resynchronization therapy (CRT) is limited by a high proportion of non-responders. Pacing activation from multiple separated left ventricular (LV) sites might improve the depolarization pattern, thereby promoting more physiological activation. To explore the effect of MPP on cardiac neuro-hormonal activity, the investigators will enroll approximately 30 patients who already underwent CRT-D implantation with a quadripolar LV lead connected to a device capable of MPP.

This pilot study will have a randomized, double-blind, cross-over design. Patients will be randomized to receive either standard biventricular pacing (MPP-OFF) or MPP (MPP-ON) within 4-6 months following the implantation procedure. Each subject will crossover to the other study group after three months. The baseline evaluation should be acquired prior to the device being programmed to the randomized setting. Repeat evaluations will be performed at the end of each 3 month crossover period.

Participation in this study will last approximately 6 months. Patients, as well as investigators other than the EP physicians, will be blinded to the pacing mode.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with a St. Jude Medical CRT-D system with MPP capability
* Patients must be willing and able to sign an appropriate informed consent form and comply with study requirements
* NT pro-BNP levels equal to or greater than 500 pg/ml.

Exclusion Criteria:

* History of stroke, PCI, myocardial infarction or unstable angina pectoris within the last 3 months.
* Atrial fibrillation with noncontrolled heart rate
* Need for intravenous inotropic support for CHF
* Classification of Status 1 for cardiac transplantation or consideration for transplantation over the next 12 months
* Undergone a cardiac transplantation
* Currently participating in any other clinical investigation
* Life expectancy < 12 months due to a disorder other than CHF
* Inability to comply with the follow-up procedures
* Patients who are or may potentially be pregnant

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Changes in blood concentrations of N-terminal pro-B type natriuretic peptide (NT pro-BNP) | Baseline. 3-Month. 6-Month.
  Changes in plasma NT pro-BNP using the difference from baseline to three months as compared to the difference from three to six months within a patient.

SECONDARY OUTCOMES:
Changes in Neurohormonal Activation | Baseline. 3-Month. 6-Month.
  Renin, Aldosteron, Norepinephrine, Endothelin-1.
Heart Failure Hospitalizations | 3-Month. 6-Month.
New York Heart Association (NYHA) Class changes | Baseline. 3-Month. 6-Month.
Changes in Quality of Life (QOL), as assessed by the Minnesota Living With Heart Failure Questionnaire | Baseline. 3-Month. 6-Month.
Echocardiographic changes | Baseline. 3-Month. 6-Month.
  Left ventricular end diastolic volume. Left ventricular end systolic volume. Left ventricular ejection fraction. Mitral regurgitation severity.
Appropriate device interventions (anti-tachycardia pacing or shock) | 3-Month. 6-Month.
Phrenic Nerve Complication Free Rate | 3-Month. 6-Month.
Occurrence of atrial and ventricular arrhythmias (amount and duration [h/day]). | 3-Month. 6-Month.
Flow-mediated vasodilation | Baseline. 3-month. 6-month
  Differences in FMD between groups
Packer's clinical composite score | Baseline. 3-month. 6-month.
  Distribution of "improved", "unchanged" and "worsened" patients as defined per Packer's clinical composite score
6-Minute-Walking-Distance | Baseline. 3 Month. 6 Month.
  The distance walked by subjects during a 6 minutes walking test

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni B Forleo, MD, PhD, Principal Investigator — University of Rome Tor Vergata
Locations (2):
- Italy (2):
  - Istituto Clinico St. Ambrogio, Milan
  - Policlinico Tor Vergata, Rome

REFERENCES:
- [Background] Pappone C, Calovic Z, Vicedomini G, Cuko A, McSpadden LC, Ryu K, Romano E, Saviano M, Baldi M, Pappone A, Ciaccio C, Giannelli L, Ionescu B, Petretta A, Vitale R, Fundaliotis A, Tavazzi L, Santinelli V. Multipoint left ventricular pacing improves acute hemodynamic response assessed with pressure-volume loops in cardiac resynchronization therapy patients. Heart Rhythm. 2014 Mar;11(3):394-401. doi: 10.1016/j.hrthm.2013.11.023. Epub 2013 Nov 28. PMID 24291411
- [Background] Rinaldi CA, Leclercq C, Kranig W, Kacet S, Betts T, Bordachar P, Gutleben KJ, Shetty A, Donal E, Keel A, Ryu K, Farazi TG, Simon M, Naqvi TZ. Improvement in acute contractility and hemodynamics with multipoint pacing via a left ventricular quadripolar pacing lead. J Interv Card Electrophysiol. 2014 Jun;40(1):75-80. doi: 10.1007/s10840-014-9891-1. Epub 2014 Mar 14. PMID 24626999